CLINICAL TRIAL: NCT03428737
Title: Impact of a Nocturnal Pressure Controlled Ventilation on Mechanical Ventilation Weaning Duration in Patients With Chronic Obstructive Respiratory Diseases REVENTIL 2
Brief Title: Impact of a Nocturnal Pressure Controlled Ventilation on Mechanical Ventilation Weaning Duration in Patients With Chronic Obstructive Respiratory Diseases
Acronym: REVENTIL 2
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: none participant included
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2017_843_0016
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Noctural Ventilatory Mode and Weaning Duration
Keywords: pressure support ventilation; pressure control ventilation; sleep, weaning; chronic obstructive respiratory disease; weaning duration period

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nocturnal controlled pressure control ventilation (Other): use of an inspiratory pressure of 20 cm of H2O and an respiratory frequency chosen to stop all spontaneous breathing activity during the night
  Interventions: Procedure: Nocturnal controlled pressure control ventilation
- Nocturnal pressure support ventilation (Other): Use of a pressure support level identical during the night to the pressure support level at the end of the day.
  Interventions: Procedure: Pressure support ventilation

INTERVENTIONS:
Procedure: Nocturnal controlled pressure control ventilation — use of an inspiratory pressure of 20 cm of H2O and an respiratory frequency chosen to stop all spontaneous breathing activity during the night
  Arms: Nocturnal controlled pressure control ventilation
Procedure: Pressure support ventilation — use of a pressure support level identical during the night to the pressure support level at the end of the day.
  Arms: Nocturnal pressure support ventilation

SUMMARY:
The weaning of mechanical ventilation is difficult period. This period is particularly difficult for patient with obstructive chronic respiratory disease and a long mechanical ventilation is associated with an increased risk of infectious complication, cardiac dysfunction, muscular weakness or barotromatism. No guideline is available on the ventilator mode to use during the night. In weaning period, some studies have demonstrated that nocturnal control ventilation during the weaning period improved the quality and the quantity of sleep. The hypothesis is that use of nocturnal controlled mechanical ventilation could decrease the weaning period duration and the ventilation weaning failure because of a sleep improvement.

The main objective is to compare mechanical ventilation weaning period duration according to the nocturnal ventilator mode (pressure controlled ventilation versus pressure support ventilation) in patients with an obstructive respiratory disease. A secondary objective is to evaluate the rate of weaning failure after the first extubation according to the nocturnal ventilator mode and to evaluate the sleep during the weaning period according to the nocturnal ventilator mode.

DETAILED DESCRIPTION:
All patients with weaning criteria, spontaneous breathing test will be done. If patient is able to have spontaneous ventilation with maximum of 16 cm of H2O of pressure support, he could be included in the study. The nocturnal ventilation mode will be randomised between pressure controlled ventilation and pressure support ventilation with the same pressure support than during the day. We will follow the quality and quantity of sleep with continue polysomnography. Indeed, patients in ICU could sleep during the night but too during the day. We will compare the duration of the weaning period between the two arms.

ELIGIBILITY:
Inclusion criteria :

* Patient with invasive mechanical ventilation (with B840 ventilator)
* Patient with ventilation weaning criteria
* Patient able to support during the day pressure support ventilation with pressure support lower than 19 cm of H2O.
* Patient with all mechanical ventilation weaning criteria for the first trial of spontaneous ventilation.
* Age > 18 years

Exclusion criteria :

* Patient with central apnoea syndrome
* Patient with narcolepsy
* Patient with metabolic encephalopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
The percentage of ventilation weaning at Day 4 | at 4 day

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Amiens, Amiens, France